CLINICAL TRIAL: NCT01216917
Title: The Influence of Ageing on Muscle Quality
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: s52701
Record Dates: First submitted 2010-10-06; First posted 2010-10-07 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2011-11

CONDITIONS: Ageing Process; Muscle Quality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Fitness
- Whole-body vibration
- Control

SUMMARY:
The purpose of the present study is to evaluate the influence of the ageing process on muscle quality. Therefore, muscle mass, muscle density and force-velocity characteristics are measured after a 5-yr interval in older adults (65+).

ELIGIBILITY:
Inclusion Criteria:

* male, +65 years
* participation in previous study "De effecten van oefenprogramma's op gezondheids- en fitheidsgerelateerde parameters in een groep van 60-plussers"
* able to perform a maximal strength test on a dynamometer

Exclusion Criteria:

* pathologies that prohibit a maximal strength test on a dynamometer

Min Age: 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: elderly men (65+)
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2010-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of kinesiology and rehabilitation sciences, Leuven, Belgium